CLINICAL TRIAL: NCT06761170
Title: Spray Cryotherapy for the Management of Benign Central Airway Stenosis (Cryo-BAS): A Randomized Controlled Trial
Brief Title: Spray Cryotherapy for the Management of Benign Central Airway Stenosis (Cryo-BAS)
Acronym: Cryo-BAS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: American Association of Broncology and Interventional Pulmonology (Unknown)
Responsible Party: Principal Investigator, Adnan Majid, MD, Chief, Section of Interventional Pulmonology, Division of Thoracic Surgery and Interventional Pulmonology, Beth Israel Deaconess Medical Center, Professor of Medicine, Harvard Medical School,, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024P000875
Record Dates: First submitted 2024-12-23; First posted 2025-01-07 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Stenosis of Trachea
Keywords: Stenosis of trachea; benign; spray cryotherapy
MeSH Terms: conditions — Tracheal Stenosis | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): 1. Stenotic lumen diameter > 8mm:
     1. Spray Cryo Therapy for 5s, repeated 3-5 cycles
     2. Balloon dilation (to normal airway diameter)
  2. Stenotic lumen diameter < 8mm
     1. Balloon dilation (up to 8mm diameter)
     2. Spray Cryo Therapy for 5s, repeated 3-5 cycles 3) Balloon dilation (to normal airway diameter)
  Interventions: Procedure: Spray cryo therapy
- Control (Active Comparator): 1. Steroid injection
  2. Radial mucosal incision
  3. Balloon dilation (to normal airway diameter)
  Interventions: Procedure: Standard of Care (SOC)

INTERVENTIONS:
Procedure: Spray cryo therapy — normal flow, 5 seconds repeated for 3-5 cycles
  Arms: Interventional
Procedure: Standard of Care (SOC) — 1. Steroid injection
  2. Radial mucosal incision
  3. Balloon dilation (to normal airway diameter)
  Arms: Control

SUMMARY:
The goal of this clinical trial is to compare spray cryotherapy plus balloon dilatation versus current standard of Care (SoC - steroid injection, radial cuts and balloon dilatation) in patients with benign airway stenosis with simple stenosis. The main question[s] investigators aim to answer are:

1. What is the need for reintervention and time to reintervention in participants with benign airway stenosis with simple stenosis who receive spray cryotherapy plus balloon dilatation versus standard of care alone?
2. To evaluate patient experience, physiological, anatomical changes, health care utilization and safety of the SCT plus balloon dilatation versus standard of care alone.

Researchers will compare spray cryotherapy plus balloon dilatation versus current standard of Care (SoC - steroid injection, radial cuts and balloon dilatation) in patients with benign airway stenosis with simple stenosis to see if it reduces the need of re intervention.

Participants will surgery and receive one of the two interventions.

DETAILED DESCRIPTION:
Investigators propose a single center, single-blinded (patient), randomized 1:1 trial comparing SCT plus Balloon dilatation (experimental group) vs SoC alone (control group). Investigators aim to recruit 50 patients.

Study will span 2-year duration with 1 year recruitment. Follow up at 6 weeks, 3 months, 6 months, 12 months. The patient's airway will be either a laryngeal mask airway or a rigid bronchoscopy for passive venting and gas egress.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with symptomatic, benign, simple stenosis of the trachea and/or subglottic space.
* 2. Stenotic airway of diameter < 1cm.

Exclusion Criteria:

1. Complex stenosis, cartilage involvement (malacia or fracture).
2. Patients with giant bullae (> a third of hemithorax) or bullae >3cm.
3. Concurrent tracheoesophageal fistula, active tracheal malignancy.
4. Presence of concomitant upper airway obstruction.
5. Pregnancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Need of re intervention | Need of re intervention in two years
  Number of patients that require new intervention for the benign airway stenosis.

SECONDARY OUTCOMES:
Time to re intervention | Two years
  Time it takes in days for a patient to need a re intervention for the benign airway stenosis after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leong P, Bardin PG, Lau KK. What's in a name? Expiratory tracheal narrowing in adults explained. Clin Radiol. 2013 Dec;68(12):1268-75. doi: 10.1016/j.crad.2013.06.017. Epub 2013 Aug 13. PMID 23953005